CLINICAL TRIAL: NCT03553823
Title: A 16-week Randomized, Open-label, Multicenter Study to Assess the Superiority of Secukinumab Over Guselkumab in the Complete Treatment of Ustekinumab Resistant Psoriatic Plaques
Brief Title: Comparison of Secukinumab Versus Guselkumab in Clearing Psoriatic Plaques Refractory to Ustekinumab
Acronym: ARROW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAIN457A2403; 2018-001048-70 (EudraCT Number)
Record Dates: First submitted 2018-05-15; First posted 2018-06-12 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Chronic Plaque-type Psoriasis
Keywords: Psoriasis; Plaque psoriasis; Secukinumab; Skin condition; skin disease; itching; psoriasis vulgaris; immune-mediated systemic disease; skin lesions; scaly patches; papules
MeSH Terms: conditions — Psoriasis; Skin Diseases; Pruritus

STUDY DESIGN:
Intervention Model Description: This was a 16-week, randomized, open-label, parallel-group, active-control study comparing secukinumab 300 mg s.c. versus guselkumab 100 mg s.c. in subjects with plaque psoriasis who had an inadequate response to ustekinumab.
Who Masked: Outcomes Assessor
Masking Description: Blinded outcome assessor assessed subjects on each visit for target plaque TCS, PASI, IGA, BSA, ppIGA, PSSI, NAPS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- secukinumab (Experimental): 20 subjects with plaque psoriasis with an inadequate response to ustekinumab self-administered 300 mg secukinumab as two 150-mg s.c. injections at Baseline, Weeks 1, 2, 3, 4 and then every 4 weeks until Week 12 inclusive
  Interventions: Procedure: Skin biopsies
- Guselkumab (Active Comparator): 20 subjects with plaque psoriasis with an inadequate response to ustekinumab self-administered guselkumab as 100 mg s.c. injections at Baseline, Weeks 4, and 12.
  Interventions: Procedure: Skin biopsies

INTERVENTIONS:
Procedure: Skin biopsies — At Baseline, two 6-mm punch biopsies were taken, one from the identified active plaque (TCS ≥ 6) and one from never-lesional skin. At the End-of-study Visit, one biopsy was taken from the same area of the active plaque sampled at Baseline.

SUMMARY:
The aim of this study was to describe the effect of direct IL-17A inhibition with secukinumab as compared with the selective inhibition of IL-23 with guselkumab (p19 subunit blocker) in controlling inflammation in psoriatic plaques that remain active despite treatment with the non-selective IL-23 inhibitor ustekinumab (blocker of p40 subunit, shared by IL-12 and IL 23).

DETAILED DESCRIPTION:
This was a 16-week, randomized, open-label, parallel-group, active-control, Phase 2a study comparing secukinumab 300 mg s.c. versus guselkumab 100 mg s.c. in subjects with plaque psoriasis who had an inadequate response to ustekinumab. Forty subjects will be randomized 1:1 and treated for 16 weeks. In each patient, a target active refractory skin plaque (TCS ≥6) is described and biopsied at baseline and at study end. The objective of the study was to assess the superiority of secukinumab over guselkumab in achieving clear/almost clear status (TCS 0-2) of the target plaques; and to describe the molecular mechanisms behind this difference

ELIGIBILITY:
Inclusion Criteria:

Chronic plaque-type psoriasis considered inadequately controlled after treatment with ustekinumab according to the following criteria-:

* Ustekinumab administered at a dose equal or higher than that on the label for at least 24 weeks. The last administration must be at least 12 weeks before randomization
* absolute PASI score of 1-10 at Screening
* Presence of at least 1 refractory skin plaque, defined by a TCS of at least 6 and severity score of at least 2 or 3 (moderate) for each individual item, with an area ≥ 10 cm2 at screening.

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and guttate psoriasis) at Screening or Baseline
* Drug-induced psoriasis (i.e., new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium) at Baseline
* Previous treatment with more than one TNFα inhibitor or with IL-17A (including secukinumab), IL-17R or IL-23 (including guselkumab) inhibitors
* Use of other investigational drugs within 4 weeks before enrolment, or within a period of 5 half lives of enrollment/initiation of the study treatment, whichever is longer
* Ongoing use of prohibited treatments (see Section 6.2.2)
* Known immunosuppression (e.g., AIDS) at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (4):
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, East Windsor, New Jersey
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Dallas, Texas
- Novartis Investigative Site, Verdun, Quebec, Canada
- Germany (9):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, Selters

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Krueger J, Langley RG, Nigen S, Kasparek T, Di Comite G, Ortmann CE, Garcet S, Kolbinger F, Reich K. Secukinumab versus guselkumab in the complete resolution of ustekinumab-resistant psoriatic plaques: The ARROW study. Exp Dermatol. 2023 Oct;32(10):1834-1847. doi: 10.1111/exd.14828. Epub 2023 Jun 5. PMID 37272375
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Screening Phase was completed by 40 (95.2%) of the 42 subjects screened. One (2.4%) subject was rescreened and 2 (4.8%) subjects failed screening
Pre-assignment Details: 39 (97.5%) subjects completed this trial
Period: Overall Study
Arm/Group | Secukinumab | Guselkumab
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Guselkumab | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 36
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.6 (15.10) | 48.5 (12.30) | 48.1 (13.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 14 | 15 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 20 | 37
  Black or African American | 2 | 0 | 2
  Asian | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Whose Plaque Achieves "Clear" or "Almost Clear" Status (TCS = 0-2)
Description: Total clinical score: number (%) of subjects who responded at Week 16 (FAS)
Time Frame: 16 week
Population: The Full Analysis Set (FAS) comprised all subjects to whom study treatment had been assigned by randomization. According to the intent-to-treat principle, subjects were analyzed according to the treatment they were assigned to during the randomization procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Guselkumab
Number analyzed (Participants) | 20 | 20
Participants | 12 | 8
Statistical Analysis 1: Comparison: Secukinumab vs Guselkumab; Proportion of subjects whose plaque achieves "clear" or "almost clear" status (TCS = 0-2); Test type: Superiority; p = 0.1715, Fisher Exact; The statistical model was the Fisher's exact test for the difference in proportions; Difference secukinumab vs guselkumab = 20.0, 95% CI 2-sided [-13.3 to 50.3]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for duration of study to week 16
Description: Adverse Events (AEs) are any untoward sign or symptom that occurs during the study treatment period
Groups:
- Secukinumab: Secukinumab
- Guselkumab: Guselkumab
Arm/Group | Secukinumab | Guselkumab
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/20
Other Adverse Events (participants affected / at risk) | 11/20 | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=20) | Guselkumab (N=20)
Gastritis (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=20) | Guselkumab (N=20)
Dacryostenosis acquired (Eye disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Gout (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Analysis of biomarkers is delayed due to the global coronavirus pandemic of 2020, thus, the biomarker-related exploratory objectives were not evaluated in this present report; but will be presented in a voluntary future update.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT03553823/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT03553823/SAP_001.pdf